CLINICAL TRIAL: NCT05920018
Title: Effects of a Combined Supplementation of Conjugated Linoleic Acid (CLA/Tonalin® FFA 80) and Probiotics (Vivomixx®/VSL#3) as add-on to a First-line Immunotherapy in Relapsing-remitting Multiple Sclerosis
Brief Title: Effects of a Combined Supplementation of Conjugated Linoleic Acid (CLA) and Probiotics (Vivomixx®) as add-on to a First-line Immunotherapy in Relapsing-remitting Multiple Sclerosis
Acronym: CLAProMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Münster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WWU21_0013
Record Dates: First submitted 2023-05-02; First posted 2023-06-27 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Linoleic Acids, Conjugated

STUDY DESIGN:
Intervention Model Description: two-arm, randomized, double-blind, placebo-controlled, multicenter
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomized after successful screening and inclusion. They will be randomized with a 1:1 ratio to receive either conjugated linoleic acid (CLA/Tonalin®) and probiotics (Vivomixx®) or the corresponding placebos as add-on therapy. Randomization will be stratified according to first-line therapy with Interferon-beta, Glatirameracetat / other glatirameroids, or Teriflunomid.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary supplement (Active Comparator): 1. Vivomixx®/VSL#3 sachets p.o. (1.800 bio bacteria/d) and
  2. Conjugated linoleic acid (CLA/Tonalin® FFA 80) capsules p.o. (2 g/d)
  Interventions: Dietary Supplement: Vivomixx®; Dietary Supplement: Conjugated linoleic acid (CLA/Tonalin® FFA 80)
- Placebo-control (Placebo Comparator): 1. Maltose as Placebo to Vivomixx® and
  2. Sunflower oil as Placebo to Conjugated linoleic acid (CLA/Tonalin® FFA 80)
  Interventions: Other: Maltose placebo; Other: Sunflower oil placebo

INTERVENTIONS:
Dietary Supplement: Vivomixx® — Daily application of four sachets, i.e. 1.800 bio bacteria/day for 48 weeks
  Arms: Dietary supplement
Dietary Supplement: Conjugated linoleic acid (CLA/Tonalin® FFA 80) — Daily application of two capsules p.o., i.e. 2g/day for 48 weeks
  Arms: Dietary supplement
Other: Maltose placebo — Daily application of four sachets for 48 weeks
  Arms: Placebo-control
Other: Sunflower oil placebo — Daily application of two capsules p.o for 48 weeks
  Arms: Placebo-control

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled multicenter study is to investigate whether the combination of food supplementation with Tonalin® and specific probiotics is a safe and effective add-on to first-line disease modifying treatment (DMT, interferon-beta derivatives as well as glatirameracetate and other glatirameroids) in relapsing remitting MS (RRMS).

100 patients will be randomly assigned in a 1:1 ratio to receive either both food supplements for 48 weeks or to receive placebo in addition to their established first-line disease modifying treatment (DMT). The two randomized groups will be compared concerning the change in volume of T2-weighted hyperintense lesions from baseline to 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting multiple sclerosis according to current McDonald Criteria, EDSS maximal 5.5, 18-60 years
* stable treatment with first-line DMT (IFNbeta, teriflunomide or glatiramer acetate/ other glatirameroids) for at least 6 months
* absence of a clinical relapse for at least 3 months before inclusion
* Written informed consent

Exclusion Criteria:

* diagnosis of primary or secondary progressive MS or other active autoimmune disease
* intake/administration of the following disease modifying therapies:

  1. at any time point: alemtuzumab, cladribine
  2. during the last 6 months before inclusion: natalizumab, fingolimod, dimethyl fumarate, siponimod
  3. during the last 12 months before inclusion: mitoxantron, ocrelizumab, ofatumumab, rituximab
* ingestion of other dietary supplementation (e.g. vitamins, probiotics, iron, calcium, prebiotics, such as omega-3-fatty acids)
* significant gastroenterological abnormality (e.g. inflammatory bowel disease, short bowel disease, preexisting digestive lesions)
* accompanying systemic immunosuppressive treatment
* relevant dietary restriction (e.g. strictly vegan nutrition)
* women during pregnancy or lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change of volume of 'hyperintense lesions in the T2-weighted MRI images' between baseline and after 48 weeks of therapy | 48 weeks
  The two randomised study groups (intervention and placebo groups) are compared with regard to the change of volume of new or enlarged 'hyperintense lesions in the T2-weighted MRI images' (hereafter T2 lesions) between the start of the study and after 48 weeks.
  T2 lesions were chosen as primary endpoint as this has been used as a surrogate marker of efficacy in several recent MS studies

SECONDARY OUTCOMES:
Change in T2 lesions at 48 weeks compared to baseline | 48 weeks
  Change in T2 lesions at 48 weeks compared to baseline (yes/no)
Number of new or enlarging T2-weighted hyperintense lesions | 48 weeks
  Number of new or enlarging T2-weighted hyperintense lesions based on the comparison of brain MRI-scans after 48 weeks of intervention as compared to baseline
Volume of new or enlarged 'hyperintense lesions in the T2-weighted MRI images' as well as double inversion recovery (DIR) images | 48 weeks
  Volume of new or enlarged 'hyperintense lesions in the T2-weighted MRI images' as well as double inversion recovery (DIR) images will be compared between the intervention arm and the placebo arm. This approach has been recently published and rises the probability to detect new brain lesions in MS without application of gadolinium with a sensitivity of 98.1%
Annualized relapse rate | 48 weeks
  All relapses confirmed by a physician will be documented and analysed. Clinical relapses are defined as onset of new or recurrent neurological symptoms lasting at least 24 hours, accompanied by objective abnormalities on a neurological examination, which are not explained solely by non-MS processes such as fever, infection, severe stress or drug toxicity. Annualized relapse rates are compared between the two study groups.

OTHER OUTCOMES:
Disease progression throughout the study | 48 weeks
  Disease progression throughout the study will be documented by assessment of the Expanded Disability Status Scale (EDSS) at baseline and at 48 weeks of the study as well as in case of unscheduled visits such as in case of a relapse. EDSS is a standardized measure of MS-related disability and a key endpoint in many clinical trials in MS.
Assessment of patient-reported outcomes (PRO) and quality of life via MSIS-29 (Multiple Sclerosis Impact Scale) | 48 weeks
  Assessment of patient-reported outcomes (PRO) and quality of life by use of the following validated and commonly used questionnaires:
  MSIS-29 (Multiple Sclerosis Impact Scale) to assess quality of life Patients will be asked to fill in this questionnaires at baseline, after 24 weeks of therapy and after 48 weeks of therapy. These additional outcomes are clinically relevant as the EDSS preferentially focuses on motor function with predominance of the lower limb.
Assessment of patient-reported outcomes (PRO) and quality of life via FSMC (Fatigue Scale for Motion and Cognition) | 48 weeks
  Assessment of patient-reported outcomes (PRO) and quality of life by use of the following validated and commonly used questionnaires:
  FSMC (Fatigue Scale for Motion and Cognition) to assess MS-related fatigue Patients will be asked to fill in this questionnaires at baseline, after 24 weeks of therapy and after 48 weeks of therapy. These additional outcomes are clinically relevant as the EDSS preferentially focuses on motor function with predominance of the lower limb.
Assessment of patient-reported outcomes (PRO) and quality of life via SDMT (Symbol-Digit Modalities Test) | 48 weeks
  Assessment of patient-reported outcomes (PRO) and quality of life by use of the following validated and commonly used questionnaires:
  SDMT (Symbol-Digit Modalities Test) to assess MS-related cognition Patients will be asked to fill in this questionnaires at baseline, after 24 weeks of therapy and after 48 weeks of therapy. These additional outcomes are clinically relevant as the EDSS preferentially focuses on motor function with predominance of the lower limb.
Assessment of patient-reported outcomes (PRO) and quality of life via HADS (Hospital Anxiety and Depression Scale) | 48 weeks
  Assessment of patient-reported outcomes (PRO) and quality of life by use of the following validated and commonly used questionnaires:
  HADS (Hospital Anxiety and Depression Scale) to assess concomitant psychiatric symptoms Patients will be asked to fill in this questionnaires at baseline, after 24 weeks of therapy and after 48 weeks of therapy. These additional outcomes are clinically relevant as the EDSS preferentially focuses on motor function with predominance of the lower limb.
Assessment of patient-reported outcomes (PRO) and quality of life via BDI-II (Beck's Depression Inventory) | 48 weeks
  Assessment of patient-reported outcomes (PRO) and quality of life by use of the following validated and commonly used questionnaires:
  BDI-II (Beck's Depression Inventory) to assess concomitant psychiatric symptoms Patients will be asked to fill in this questionnaires at baseline, after 24 weeks of therapy and after 48 weeks of therapy. These additional outcomes are clinically relevant as the EDSS preferentially focuses on motor function with predominance of the lower limb.
Assessment of patient-reported outcomes (PRO) and quality of life via TSQM-9 (Treatment Satisfaction Questionnaire for Medication) | 48 weeks
  Assessment of patient-reported outcomes (PRO) and quality of life by use of the following validated and commonly used questionnaires:
  TSQM-9 (Treatment Satisfaction Questionnaire for Medication) to assess treatment satisfaction Patients will be asked to fill in this questionnaires at baseline, after 24 weeks of therapy and after 48 weeks of therapy. These additional outcomes are clinically relevant as the EDSS preferentially focuses on motor function with predominance of the lower limb.
Changes in key peripheral blood immune signatures | 48 weeks
  Highly standardized flow-cytometry of PBMC will be performed in order to determine treatment-related changes in peripheral immune signatures.
Focus on signs of gastrointestinal and systemic side effects | 48 weeks
  The rate and nature of adverse events, changes in vital signs and physical examinations, and abnormal laboratory results will be documented and analysed.
Functional characterization of human myeloid cells | 48 weeks
  A comprehensive and detailed characterization of all major immune cell populations of the peripheral blood will be done. In addition a characterization of their maturity status, their activation state, as well as certain functional properties including cytokine production as well as production of cytolytic molecules will be assessed. The aim of the immunological analysis of peripheral blood immune signatures is to investigate whether a change in the composition and activation state of the immune cells in the peripheral blood can be observed as a consequence of the combined intervention with Tonalin® and Vivomixx® as compared to the placebo group. A particular focus will be on the reduction in proinflammatory properties of different myeloid cell populations, based on our preliminary work. The different immune cell populations will be analyzed both as percentages and as absolute cell numbers.
Correlation of identified immunological effects with main endpoints of MRI and clinical efficacy | 48 weeks
  The correlation of identified immunological effects with main endpoints of MRI (including rate of global brain and grey matter atrophy derived from structural MRI) and clinical efficacy will be analysed using multivariable regression methods or machine learning approaches.
Changes in diffuse white matter damage (measured by fractional anisotropy FA) | 48 weeks
  Changes in diffuse white matter damage (measured by fractional anisotropy FA)
Global brain atrophy, grey matter atrophy and white matter atrophy | 48 weeks
  Rate of global brain and grey matter atrophy derived from structural MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Klotz, Prof., Principal Investigator — Universität Münster
Locations (4):
- Germany (4):
  - Universitätsklinik Heidelberg, Neurologische Klinik, Heidelberg, Baden-Wurttemberg
  - Neurological study centre, Department of Neurology, Mainz, Hesse
  - IIT unit of the Department of Neurology with Institute of Translational Neurology, Münster, North Rhine-Westphalia
  - Klinikum Osnabrück GmbH, Klinik für Neurologie, Osnabrück, North Rhine-Westphalia